Alcon - Business Use Only Protocol - Clinical Effective Document: TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT Effective Date: 01-Mar-2018

Document: TDOC-0054838 Status: Effective 



Title:

# **Clinical Evaluation of Two Monthly Contact Lenses**

| Protocol Number: | CLD523-E001/ NCT03459131 | |
|---|---|---|
| Sponsor Name and Address: | Alcon Research, Ltd.<br>6201 South Freeway<br>Fort Worth, Texas 76134-2099 | |
| Test Product(s): | Biofinity® Energys <sup>TM</sup> contact lenses | |
| Investigator Agreement: | I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practice (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Additionally, I will comply with all procedures for data recording and reporting, will permit monitoring, auditing, and inspection of my research center, and will retain all records until notified by the Sponsor. | |
| Principal Investigator: | | |
| | Signature | Date |
| Name: | | |
| Address: | | |

Effective Date: 01-Mar-2018

Alcon - Business Use Only Protocol - Clinical Effective Document: TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT

Document: TDOC-0054838 Status: Effective 

## 1 PROTOCOL SYNOPSIS

| Trial Sponsor | Alcon Research, Ltd. |
|---|---|
| _ | 6201 South Freeway |
| | Fort Worth, Texas 76134-2099 |
| Name of Test Product(s) | CooperVision® BIOFINITY ENERGYS soft contact lenses |
| | (BIOFINITY ENERGYS) |
| Name of Control | Cooper Vision BIOFINITY soft contact lenses (BIOFINITY) |
| Product(s) | |
| Title of Trial | Clinical Evaluation of Two Monthly Contact Lenses |
| Protocol Number | CLD523-E001 |
| Number of Sites | 1 |
| Country | US |
| Planned Duration of | Up to 18 days total duration |
| Exposure | Test Product: 7 days (±2 days) |
| | Control Product: 7 days (± 2 days) |
| Number of Subjects | Target to complete: 10 |
| | Planned to enroll: ~16 |
| Study Population | Volunteer subjects aged 18 to 35 with normal eyes (other |
| | than correction for refractive error), currently wearing |
| | BIOFINITY (or private label) sphere soft contact lenses on a |
| | daily wear basis. Subjects should have at least 3 months of |
| | BIOFINITY (or private label) wearing experience, wear |
| | these lenses at least 5 days per week and at least 8 hours per |
| | day, use digital devices at least 4 hours per day at least 5 |
| | days per week, and require contact lenses in a power range |
| | from +6.00 to -10.00 DS. |
| Objective(s) | The primary objective is to explore overall vision with BIOFINITY ENERGYS as compared to BIOFINITY lenses after 1 week of wear. |
| | The secondary objective is to evaluate the difference in over-<br>refraction of BIOFINITY ENERGYS as compared to<br>BIOFINITY. |
| Endpoints | Primary Effectiveness |
| | Overall Vision |
| | Secondary Effectiveness |
| | Over-refraction |

Document: TDOC-0054838
Status: Effective 

| | Safety |
|---|---|
| | • AEs |
| | Biomicroscopy findings |
| Assessments | Device deficiencies Effectiveness |
| T is substitution of the s | <ul> <li>VA with study lenses (OD, OS, OU / Snellen, Distance)</li> <li>Manifest refraction</li> <li>BCVA (Snellen distance with manifest refraction)</li> <li>Over refraction with study lenses</li> </ul> |

Effective Date: 01-Mar-2018 Alcon - Business Use Only Protocol - Clinical Effective

Document: TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT

Document: TDOC-0054838
Status: Effective 

| Status: Effective | | 1 age 4 01 40 |
|---|---|---|
| | Safety • AEs | |
| | Biomicroscopy Device deficiencie | |
| Ctudu Davian | | |
| Study Design | | ☐ Single-masked (trial subject) ☐ Single-masked (Investigator) ☑ Double-masked ☐ Open-label ☐ Other |
| | ☐ Contralateral ☐ Bilateral ☐ Monocular lens wear | Randomized |
| Test Product 1 Details | Primary component/material | comfilcon A |
| | Product Name | BIOFINITY ENERGYS |
| | LID Number | NA |
| | Manufacturer | CooperVision |
| | Other | +6.00 DS to -6.00 DS (0.25 steps)<br>-6.50 DS to -10.00 DS (0.50 steps) |
| Control Product Details | Primary component/material | comfilcon A |
| | Product Name | BIOFINITY |
| | LID Number | NA |
| | Manufacturer | CooperVision |
| | Other | +6.00 DS to -6.00 DS (0.25 steps)<br>-6.50 DS to -10.00 DS (0.50 steps) |
| Inclusion Criteria | <ol> <li>Subject must be 18 to</li> <li>Subject must be able</li> </ol> | 35 years of age. to understand and must sign an ICF |

Effective Date: 01-Mar-2018

Alcon - Business Use Only Protocol - Clinical Effective Document; TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT Status: Effective Page **5** of **43** 

| | | 6 |
|---|---|---|
| | | that has been approved by an IRB. |
| | 3. | Successful wear of BIOFINITY (spherical) (or private |
| | | label) contact lenses in both eyes for a minimum of 5 |
| | | days per week and 8 hours per day during the past 3 |
| | | months. |
| | 4. | Manifest cylinder $\leq 0.75$ D in each eye. |
| | 5. | BCVA 20/25 or better in each eye. |
| | 6. | Subject must possess spectacles that provide a corrected |
| | | VA of 20/40 or better OU and be willing to wear them |
| | | (as needed). |
| | 7. | Currently using digital devices (computer, tablet, and/or |
| | | smart phone) for a minimum of 5 days per week and 4 |
| | | hours per day. |
| Exclusion Criteria | 1. | Any anterior segment infection, inflammation, or |
| | | abnormality or disease (including systemic) that |
| | | contraindicates contact lens wear, as determined by the |
| | | Investigator. |
| | 2. | Any use of systemic or ocular medications for which |
| | | contact lens wear could be contraindicated, as |
| | | determined by the Investigator. |
| | 3. | History of refractive surgery or plan to have refractive |
| | | surgery during the study or irregular cornea in either eye. |
| | 4. | Ocular or intraocular surgery (excluding placement of |
| | | punctal plugs) within the previous 12 months or planned |
| | | during the study. |
| | 5. | Biomicroscopy findings at screening that are moderate |
| | | (Grade 3) or higher and/or corneal vascularization that is |
| | | mild (Grade 2) or higher. |
| | 6. | Current or history of pathologically dry eye in either eye |
| | | that, in the opinion of the Investigator, would preclude |
| | | contact lens wear. |
| | 7. | Current or history of herpetic keratitis in either eye. |
| | 8. | Eye injury in either eye within 12 weeks immediately |
| | | prior to enrollment for this trial. |
| | 9. | Current or history of intolerance, hypersensitivity or |
| | | allergy to any component of the study products. |
| | 10 | . Wearing habitual contact lenses in an extended wear |

Effective Date: 01-Mar-2018 Alcon - Business Use Only Protocol - Clinical Effective Document: TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT

Document: TDOC-0054838 Status: Effective 

| | modality (routinely sleeping in lenses for at least 1 night |
|---|---|
| | per week) over the last 3 months prior to enrollment. |
| | 11. Any use of topical ocular medications that would require |
| | instillation during contact lens wear. |
| | 12. The Investigator, his/her staff, family members of the |
| | Investigator, family members of the Investigator's staff, |
| | or individuals living in the households of the |
| | aforementioned persons may not participate in the study. |
| | 13. Participation of the subject in a clinical trial within the |
| | previous 30 days or currently enrolled in any clinical |
| | trial. |
| Associated Materials | Lenses will be cared for with subject's habitual lens care solution. |
| | Use of habitual lubricating/re-wetting drops will be |
| | permitted during the trial. |
| | permitted during the trial. |
| | If study lenses are not available for dispensing at Visit 2, use |
| | of habitual lenses will be permitted between Visits 1 and 2, |
| | up to 7 days, before dispensing of study lenses. |
| | up to 7 days, before dispensing of study lenses. |

Table 1-1 Schedule of Study Procedures and Assessments

| | | | Visit 2 | Vis | it 3 | Visit 4 | sit | |
|---|---|---|---|---|---|---|---|---|
| Procedure/ Assessment | | Visit 1 | 0-7 days<br>from V1 | | days<br>V2 | 7 (±2) days<br>from V3 | ed Visit | Exit |
| | Pre-screening | Baseline /<br>Fitting | Dispense<br>Pair 1 | Follow-up<br>Pair 1 | Dispense<br>Pair 2 | Follow-up<br>Pair 2 /<br>Exit | Unscheduled | Early Exit |
| Digital Use Time | <b>√</b> ∗ | | | ✓ | | ✓ | ✓ | ✓ |
| Informed Consent | | ✓ | | | | | | |
| Demographics | | ✓ | | | | | | |
| Medical History | | ✓ | ✓ | ✓ | | ✓ | ✓ | ✓ |
| Concomitant Medications | | ✓ | (✓) | (✓) | | (√) | (√) | (✓) |
| Inclusion/Exclusion | | ✓ | | | | | | |


Status: Effective 

| Servers. | | | | | | | age / c | |
|---|---|---|---|---|---|---|---|---|
| Procedure/ Assessment | ng | Visit 1 | Visit 2 0-7 days | | it 3<br>) days | Visit 4 7 (±2) days | Visit | ţ |
| | eni | | from V1 | fron | n V2 | from V3 | ed | Exi |
| | Pre-screening | Baseline /<br>Fitting | Dispense<br>Pair 1 | Follow-up<br>Pair 1 | Dispense<br>Pair 2 | Follow-up<br>Pair 2 /<br>Exit | Unscheduled Visit | Early Exit |
| Habitual lens* (brand, power) / Lens care* (brand) / Rewetting drops* (Brand / usage) | | <b>√</b> | | | | | | |
| Manifest refraction* | | ✓ | (✓) | (* | <b>(</b> ) | (✓) | <b>(√)</b> | (✓) |
| BCVA (OD, OS, Snellen<br>distance with manifest<br>refraction) * | | ✓ | (✓) | (* | <b>(</b> ) | (✔) | <b>(√)</b> | <b>(</b> ✓) |
| Biomicroscopy | | ✓ | ✓ | ✓ | | ✓ | ✓ | ✓ |
| Dispense study lenses / Rx | | | ✓ | | ✓ | | | |
| Over-refraction (OD, OS) | | | ✓ | | ✓ | | | |
| VA w/ study lenses (OD, OS, OU, Snellen distance,) | | | ✓ | <b>✓</b> | <b>✓</b> | ✓ | <b>(√)</b> | <b>√</b> |
| AEs | | ✓ | ✓ | v | / | ✓ | ✓ | ✓ |
| Device deficiencies | | ✓ | ✓ | • | | ✓ | <b>✓</b> | ✓ |
| Exit Form | | (✓) | (✓) | (, | <u>()</u> | (✓) | <b>(√)</b> | ✓ |

<sup>(✓)</sup> assessment performed as necessary, eg, decrease of VA by 2 lines or more with investigational product (IP)

<sup>\*</sup> Source only

Effective Date: 01-Mar-2018

Alcon - Business Use Only Protocol - Clinical Effective Document: TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT Status: Effective 

## 1.1 Abbreviations

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| CFR | Code of Federal Regulations |
| eCRF | Electronic case report form |
| DS | Diopter sphere |
| EDC | Electronic data capture |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| ISO | International Organization for Standardization |
| LID | Lens identification |
| mm | Millimeter |
| MOP | Manual of procedures |
| NA | Not applicable |
| OD | Right eye |
| OS | Left eye |
| OU | Both eyes |
| Rx | Prescription |
| SAE | Serious adverse event |
| SADE | Serious adverse device effect |
| US | United States |
| VA | Visual acuity |

| Do | lcon - Bus<br>ocument: TDO<br>atus: Effect | C-0054838 | Protocol - Clinical Version: 2.0; Most-Recent; Effective; | Effective Date: 01-Mar-2018 CURRENT |
|---|---|---|---|---|
| 2 | TABLE | OF CONTE | NTS | |
| Cl | inical Eval | uation of Two N | Ionthly Contact Lenses | 1 |
| 1 | PROTOG | COL SYNOPSIS | | 2 |
| | 1.1 | Abbreviations | | 8 |
| 2 | TABLE ( | OF CONTENTS | | 9 |
| Lis | st of Table | S | | 11 |
| Lis | st of Figur | es | | 11 |
| 3 | INTROD | UCTION | | 12 |
| | 3.1 | Study Rational | e and Purpose | 12 |
| | 3.2 | • | | |
| | 3.3 | Risks and Bene | fits | 12 |
| | 3.4 | Subject Popula | tion | 13 |
| | 3.5 | Outline of Stud | у | 13 |
| 4 | TREATM | MENTS ADMIN | ISTERED | 14 |
| | 4.1 | Identity of Stud | ly Treatments | 14 |
| | 4.2 | Accountability | Procedures | 15 |
| | 4.3 | Local Lens Pro | curement | 16 |
| | | 4.3.1 Proce | rement | 16 |
| | | 4.3.2 Labe | ing | 16 |
| | | | ling | |
| | | - | ensing and Accountability | |
| | | | Disposition | |
| | 4.4 | | lection, Storage and Return | |
| 5 | STUDY | PROCEDURES | AND ASSESSMENTS | 17 |
| | 5.1 | | ninations | |
| | | | 1 (Day 0) – Baseline/Fitting | |
| | | | 2 (0-7 Days from Visit 1) – Dispense Pa | |
| | | | $3 (7 \pm 2 \text{ Days from Visit 2}) - [Follow-upensing visit for Pair 2]$ | |
| | | - | 4 (7 $\pm$ 2 Days from Visit 3) – [Follow-up | |
| | 5.2 | Unscheduled V | isits | 24 |
| | 5.3 | Discontinued S | ubjects | 25 |

Printed By:

| | con - Bus | mess ese emj | te: 01-Mar-2018 |
|---|---|---|---|
| Sta | atus: Effect | | |
| | 5.4 | Clinical Study Termination | 25 |
| 6 | ANALYS | SIS PLAN | 26 |
| | 6.1 | Subject Evaluability | 26 |
| | 6.2 | Analysis Data Sets | 26 |
| | | 6.2.1 Safety Analysis Set | 26 |
| | 6.3 | Demographic and Baseline Characteristics | 27 |
| | 6.4 | Effectiveness Analyses | 27 |
| | | 6.4.1 Primary Effectiveness | 27 |
| | | 6.4.1.1 Statistical Hypotheses | 27 |
| | | 6.4.1.2 Analysis Methods | |
| | | 6.4.2 Secondary Effectiveness | 27 |
| | | 6.4.2.1 Statistical Hypotheses | 27 |
| | | 6.4.2.2 Analysis Methods | |
| | | | 28 |
| | | | 28 |
| | . <b>.</b> | | 28 |
| | 6.5 | Subgroup Analyses | |
| | 6.6 | Handling of Missing Data | |
| | 6.7 | Multiplicity | 29 |
| | 6.8 | Safety Analysis | 29 |
| | 6.9 | Interim Analyses | 29 |
| | 6.10 | Sample Size Justification | 30 |
| 7 | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 30 |
| | 7.1 | General Information | 32 |
| | 7.2 | Monitoring for Adverse Events | 35 |
| | 7.3 | Procedures for Recording and Reporting | 35 |
| | 7.4 | Return product analysis | 37 |
| | 7.5 | Follow-Up of Subjects with Adverse Events | 37 |
| | 7.6 | Pregnancy in the Clinical Study | 38 |
| 8 | CONFID | ENTIALITY, BIAS, AND MASKING | 38 |
| | 8.1 | Subject Confidentiality and Methods Used to Minimize Bias | 38 |
| | 8.2 | Unmasking of the Study Treatment | |
| 9 | DATA H | ANDLING AND ADMINISTRATIVE REQUIREMENTS | |

| | iness ese only | ate: 01-Mar-2018 |
|---|---|---|
| Document: TDO Status: Effect | | |
| 9.1 | Completion of Source Documents and Case Report Forms | 39 |
| 9.2 | Data Review and Clarifications | 40 |
| 9.3 | Regulatory Documentation and Records Retention | 40 |
| 10 ETHICS | AND COMPLIANCE | 40 |
| 10.1 | Compliance | 41 |
| 10.2 | Institutional Review Board (IRB) | 41 |
| 11 PROTOG | COL AMENDMENT HISTORY | 42 |
| 12 REFERE | ENCES | 43 |
| 12.1 | References applicable for all clinical trials | 43 |
| | 12.1.1 US references applicable for clinical trials | 43 |
| 12.2 | References for this clinical trial | 43 |
| Table 1-1 | List of Tables Schedule of Study Procedures and Assessments | 6 |
| | List of Figures | |
| Figure 7–1 | Categorization of All AEs | 32 |
| Figure 7-2 | Categorization of All Serious Adverse Events | 33 |


Status: Effective 

#### 3 INTRODUCTION

## 3.1 Study Rationale and Purpose

The purpose of this study is to obtain on-eye performance data to aid contact lens product development. The primary and secondary endpoints were selected to fulfil the primary and secondary objectives of the study. Procedures for measurement of these endpoints were selected based on common practice for these assessments. The design of this study is justified based upon FDA approval and information, as described within the Package Inserts. BIOFINITY contact lenses were chosen as the control product because these lenses have the same wear modality, material, and parameters to the test product BIOFINITY ENERGYS, and are the spherical design as compared to the aspherical design, respectively.

There are no immediate plans to submit the results of this early clinical development study for publication; however, the results may be offered for publication if they are of scientific interest, or if the results relate to a product that is subsequently approved or cleared for marketing.

## 3.2 Trial Objective

The primary objective is to explore overall vision with BIOFINITY ENERGYS as compared to BIOFINITY lenses after 1 week of wear.

The secondary objective is to evaluate the difference in over-refraction of BIOFINITY ENERGYS as compared to BIOFINITY.

#### 3.3 Risks and Benefits

Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. Material properties and design characteristics of the contact lens in development are features consistent with successful contact lens wear.

Both study contact lens are for daily wear use under a weekly/monthly wear modality. A summary of the known potential risks and benefits associated with these marketed contact lenses can be found in the package inserts, See MOP. Risks are minimized by compliance with the eligibility criteria and study procedures, and through close supervision by a licensed clinician during exposure to the study lenses. In general, the risks with the marketed contact lenses in this study are anticipated to be similar to other marketed weekly/monthly soft contact lenses.


Status: Effective 

The site personnel will educate subjects on proper hygiene and lens handling, and compliance with the use of contact lenses according to the protocol. Subjects should be instructed not to wear contact lenses while sleeping or swimming. The site personnel will also advise the subjects to remove contact lenses and return for prompt follow-up of symptoms, such as ocular discomfort, foreign body sensation, excessive tearing, vision changes, or hyperemia.

## 3.4 Subject Population

The study population includes approximately 16 volunteer subjects to be enrolled at 1 site. The study population will consist of subjects aged 18 to 35 with normal eyes (other than correction for refractive error), currently wearing BIOFINITY sphere soft contact lenses (or private label) on a daily wear basis. Subjects should have at least 3 months of BIOFINITY (or private label) wearing experience, wear these lenses at least 5 days per week and at least 8 hours per day, use digital devices at least 4 hours per day at least 5 days per week, and require contact lenses in a power range from +6.00 to -10.00 DS.

Subjects must be screened according to the full list of inclusion/exclusion criteria in Section 1 of this protocol.

After informed consent is signed, a separate screening visit is allowed for the following criteria:

- INC01 Subject must be 18 to 35 years of age
- EXC13 Participation of the subject in a clinical trial within the previous 30 days or currently enrolled in any clinical trial

This separate screening visit can take place regardless of whether any other criterion has been verified.

Rescreening of subjects is not allowed in this study.

#### 3.5 Outline of Study

This will be a single-site, prospective, randomized, double-masked, bilateral crossover study comparing 2 weekly/monthly contact lenses. The expected duration of subject participation in the study is  $7 \pm 2$  days per lens type, with up to 4 scheduled visits. The study is expected to be completed in approximately 4 weeks.


Status: Effective 

## 4 TREATMENTS ADMINISTERED

Subjects will be randomized in a 1:1 manner to receive treatment in crossover sequence, BIOFINITY ENERGYS then BIOFINITY, or BIOFINITY then BIOFINITY ENERGYS, respectively.

# 4.1 Identity of Study Treatments

| DESCRIPTION OF TEST AND CONTROL PRODUCTS | | |
|---|---|---|
| | Test Product | Control Product |
| Lens identified in randomization system as: | BIOFINITY ENERGYS | BIOFINITY |
| Lens | BIOFINITY ENERGYS | BIOFINITY |
| Material | comfilcon A | comfilcon A |
| Water Content | 48% | 48% |
| Base Curve (mm) | 8.6 | 8.6 |
| Diameter (mm) | 14.0 | 14.0 |
| Rx powers to be available in this study | +6.00 DS to -6.00 DS (0.25 steps)<br>-6.50 DS to -10.00 DS (0.50 steps) | +6.00 DS to -6.00 DS (0.25 steps)<br>-6.50 DS to -10.00 DS (0.50 steps) |
| Packaging, Labeling, and Supply | Blister foil pack in commercial packaging Foil label includes at a minimum: material name base curve diameter packing solution power lot number expiration date content statement Manufacturer information country of origin. Site will procure study lenses locally. Lenses should be stored at room temperature. | Blister foil pack in commercial packaging Foil label includes at a minimum: material name base curve diameter packing solution power lot number expiration date content statement Manufacturer information country of origin Site will procure study lenses locally. Lenses should be stored at room temperature. |


Status: Effective 

| Usage | • Wear: |
|-------|-----------------------------------------------------------------|
| | o Daily Wear |
| | <ul> <li>Bilateral Crossover</li> </ul> |
| | • Replacement period: Not applicable for $7 \pm 2$ days of wear |
| | with these monthly lenses. Replacement lenses will not be |
| | provided to the subjects. In the event a lens needs to be |
| | replaced, the subject must return to the site for a replacement |
| | lens. |
| | Exposure: Up to 18 days total duration |
| | <ul> <li>Test Product: 7 days (± 2 days)</li> </ul> |
| | <ul> <li>Control Product: 7 days (± 2 days)</li> </ul> |
| | Lens Care: Cleaned and disinfected with subject's habitual lens |
| | care solution after each use |
| | Instructions for use are provided in the MOP |

## 4.2 Accountability Procedures

Upon receipt of the study lenses, the Investigator or delegate will conduct an inventory. Designated unmasked study staff will provide the study lenses to the subjects in accordance with their randomization schedule. Throughout the study, the Investigator or delegate must maintain records of study treatment dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of clinical supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation.

It is the Investigator's responsibility to ensure that:

- · All study products are accounted for and not used in any unauthorized manner
- All used foils and unused supplies are returned by each subject
- All unused products are available for return to the Study Sponsor, as directed
- Any study lenses associated with a device deficiency or with any product-related adverse
  event [ie, ADE or SADE], that are related to comfort or vision, are returned to the Study
  Sponsor for investigation. Refer to MOP of this protocol for additional information on the
  reporting of device deficiencies and AEs and the return of study products associated with
  these events.


Status: Effective 

#### 4.3 Local Lens Procurement

Site will procure all study lenses locally and the following procedures are to be followed.

#### 4.3.1 Procurement

Site will procure commercial lenses through their standard channels. The site must follow any recalls from the distributor/manufacturer for locally procured lenses. Site personnel dispensing lenses must ensure the contact lenses being dispensed are not expired.

## 4.3.2 Labeling

All study lenses will be provided to subject in commercial packaging.

## 4.3.3 Handling

Lenses will be stored in a safe, secure location with limited access and separated from general stock. Designated site staff should follow the manufacturer's instructions on the storage requirements of the lenses.

## 4.3.4 Dispensing and Accountability

Lenses are to be provided to the subjects in accordance with Protocol. The Investigator or delegate is to maintain records of the dispensation and collection of all study lenses. This record will be made available to the Sponsor's monitor to account for all study lenses.

It is the Investigator's responsibility to ensure that all used study lens lidding foils dispensed to each subject are saved, and that they are available for the clinical study monitor to perform final accountability. Any discrepancy and/or deficiency must be recorded, with an explanation.

## 4.3.5 Final Disposition

At the conclusion of the study, once the Clinical Study Manager has performed a final reconciliation of the accountability records, unused study lenses reimbursed by the Sponsor will be returned to the Sponsor.


Status: Effective 

## 4.4 Worn Lens Collection, Storage and Return

See MOP for instructions on lens storage and return.

#### 5 STUDY PROCEDURES AND ASSESSMENTS

## 5.1 Visits and Examinations

Detailed descriptions of assessments and procedures are provided below. The Investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

## 5.1.1 Visit 1 (Day 0) – Baseline/Fitting

| 1 | Explain the purpose and nature of the study, and have the subject read, sign, and date |
|---|---|
| | the IRB-approved informed consent document. Additionally, have the individual |
| | obtaining consent from the subject and a witness, if applicable, sign and date the |
| | informed consent document. Provide a photocopy of the signed document to the |
| | subject and place the original signed document in the subject's chart. After signing |
| | the ICF, a subject will be assigned a subject number by the EDC system. A signed |
| | informed consent document defines the point of enrollment. |
| 2 | Obtain demographic information and medical history, including information on all |
| | medications used within the past 30 days. Include herbal therapies, vitamins, and all |
| | over-the-counter as well as prescription medications. |
| 3 | Record habitual lens information (brand, power)*, lens care information (brand)*, |
| | and re-wetting drops (brand / usage).* |
| | *Source only |
| 4 | Perform a manifest refraction.* |
| | *Source only |
| 5 | Perform Snellen BCVA with manifest refraction.* |
| | OD & OS, distance only |
| | Note: Distance BCVA must be 20/25 or better in each eye for the subject to qualify for the |
| | study. *Source only. |


Status: Effective 

| 6 | Perform slit-lamp biomicroscopy (without contact lenses) to evaluate the following: |
|---|---|
| | Limbal hyperemia |
| | Bulbar hyperemia |
| | Corneal staining |
| | Conjunctival staining |
| | Palpebral conjunctival observations |
| | Corneal epithelial edema |
| | Corneal stromal edema |
| | Corneal vascularization |
| | Conjunctival compression/indention |
| | Chemosis |
| | Corneal infiltrates |
| | Other findings |
| 7 | Determine study lens powers based upon the manifest refraction and habitual lens |
| | powers. |
| 8 | Review inclusion/exclusion criteria to determine if the subject qualifies to be |
| | randomized into the study. If subject qualifies, request randomization. If subject does |
| | not qualify, exit the subject from the study as a screen failure. |
| 10 | Assess and record any AEs and device deficiencies reported or observed during the |
| | study visit. |
| | Note: AEs and device deficiencies must be recorded for all enrolled subjects from the time of |
| | signature of informed consent including those that screen fail. |
| 11 | If study lens powers have not changed from habitual Rx, then can use study lenses |
| | ordered after Pre-screening and proceed with Visit 2. |
| | Note: Visit 2 may occur on same day as Visit 1 when lenses do not have to be re-ordered. |
| 12 | If study lens powers have changed, then study lenses must be re-ordered. Schedule |
| | Visit 2 to take place 0-7 days after Visit 1. |

# 5.1.2 Visit 2 (0-7 Days from Visit 1) – Dispense Pair 1

| 1 | If Visit 2 occurs on same day as Visit 1, go to line 5 of this visit. |
|---|---|
| | Obtain information on any changes in medical health and/or the use of concomitant |
| | medications. |

Alcon - Business Use Only Protocol - Clinical Effective Document: TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT Effective Date: 01-Mar-2018

Document: TDOC-0054838 Status: Effective 

| 2 | Record any device deficiencies or AEs including those associated with changes in |
|---|---|
| | concomitant medication dosing, which are observed or reported since the previous |
| | visit. |
| 3 | Perform Snellen BCVA with manifest refraction.* (as necessary). |
| | OD & OS, distance only |
| | • OD & OS, distance only |
| | Note: Perform only as necessary, ie, decrease of VA by 2 lines or more with IP. |
| | *Source only. |
| 4 | Perform slit-lamp biomicroscopy (without contact lenses) to evaluate the following: |
| | Limbal hyperemia |
| | Bulbar hyperemia |
| | Corneal staining |
| | Conjunctival staining |
| | <ul> <li>Palpebral conjunctival observations</li> </ul> |
| | Corneal epithelial edema |
| | Corneal stromal edema |
| | Corneal vascularization |
| | Conjunctival compression/indention |
| | <ul><li>Chemosis</li><li>Corneal infiltrates</li></ul> |
| | Other findings |
| 5 | Dispense Pair 1 study lenses. Provide the subject with written and verbal |
| | instructions on lens wear and habitual lens care. |
| 6 | Based upon the randomized treatment sequence assignment, have the subject insert |
| | the Pair 1 study lenses. |
| | <ul> <li>Keep all lidding foils of lenses for study lens accountability.</li> </ul> |
| | Follow procedures to maintain masking. |
| 7 | Evaluate Pair 1 study lenses by performing the following: |
| | <ul> <li>Snellen VA with study lenses, without over-refraction (OD, OS, OU at</li> </ul> |
| | distance)* |
| | Over-refraction to determine the best contact lens-corrected VA |
| | *VA w/study lenses must be 20/40 OU or better for subject to leave the office |
| | 1 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 |


Status: Effective 



# 5.1.3 Visit 3 (7 ± 2 Days from Visit 2) – [Follow-up visit for Pair 1 and Dispensing visit for Pair 2]

- Obtain information on any changes in medical health and/or the use of concomitant medications.

  Record any device deficiencies or AEs including those associated with changes in concomitant medication dosing, which are observed or reported since the previous visit(s).
- 3 Review subject compliance with lens wear and adjunct product usage.
- 5 Perform Snellen BCVA with manifest refraction.\* (as necessary).
  - OD & OS, distance only

**Note: Perform only as necessary**, ie, decrease of VA by 2 lines or more with IP. \*Source only.

Effective Date: 01-Mar-2018 

Document: TDOC-0054838
Status: Effective 

| 6 | Evaluate Pair 1 study lenses by performing the following: |
|---|---|
| | • Snellen VA with study lenses (OD, OS, OU at distance) |
| 8 | Perform slit-lamp biomicroscopy (without contact lenses) to evaluate the following: |
| | <ul> <li>Limbal hyperemia</li> <li>Bulbar hyperemia</li> <li>Corneal staining</li> <li>Conjunctival staining</li> <li>Palpebral conjunctival observations</li> <li>Corneal epithelial edema</li> <li>Corneal stromal edema</li> <li>Corneal vascularization</li> <li>Conjunctival compression/indention</li> <li>Chemosis</li> <li>Corneal infiltrates</li> <li>Other findings</li> </ul> |
| 10 | Dispense Pair 2 study lenses. Provide the subject with written and verbal |
| | instructions on lens wear and habitual lens care. |


Status: Effective 

| | · |
|---|---|
| 11 | Evaluate Pair 2 study lenses by performing the following: |
| | Snellen VA with study lenses, without over-refraction (OD, OS, OU at |
| | distance)* |
| | Over-refraction to determine the best contact lens-corrected VA |
| | *VA w/study lenses must be 20/40 OU or better for subject to leave the office |
| 13 | Assess and record any AEs and device deficiencies reported or observed during the |
| | study visit. |
| | Note: AEs and device deficiencies must be recorded for all enrolled subjects from the time |
| | of signature of informed consent including those that screen fail. |
| 14 | Schedule Visit 4 to take place $7 \pm 2$ days after Visit 3. |
| 15 | Note: If for some reason a subject is unable to wear a study lens for the duration of |
| | this visit window, instruct the subject to return to the site for an Unscheduled Visit |
| | as well as lens removal on site, if possible. If study lenses need to be replaced, |
| | unmasked study personnel may do so at this visit The subject should then be |
| | scheduled to return to the clinic for Visit 4 (if possible) or exited from the study. |

# 5.1.4 Visit 4 (7 $\pm$ 2 Days from Visit 3) – [Follow-up visit for Pair 2 / Exit]

| 1 | Obtain information on any changes in medical health and/or the use of concomitant medications. |
|---|---|
| 2 | Record any device deficiencies or AEs including those associated with changes in concomitant medication dosing, which are observed or reported since the previous visit(s). |
| 3 | Review subject compliance with lens wear and adjunct product usage. |
| 3 | Review subject compliance with lens wear and adjunct product usage. |

Effective Date: 01-Mar-2018 

Document: TDOC-0054838
Status: Effective 

| 5 | Perform Snellen BCVA with manifest refraction.* (as necessary). |
|---|---|
| | OD & OS, distance only |
| | Note: Perform only as necessary, ie, decrease of VA by 2 lines or more with IP. |
| | *Source only. |
| 6 | Evaluate Pair 2 study lenses by performing the following: |
| | <ul> <li>Snellen VA with study lenses (OD, OS, OU at distance)</li> </ul> |
| 8 | Perform slit-lamp biomicroscopy (without contact lenses) to evaluate the following: |
| | Limbal hyperemia |
| | Bulbar hyperemia |
| | Corneal staining |
| | Conjunctival staining |
| | Palpebral conjunctival observations |
| | Corneal epithelial edema |
| | Corneal stromal edema |
| | Corneal vascularization |
| | Conjunctival compression/indention |
| | Chemosis |
| | Corneal infiltrates |
| | Other findings |


Status: Effective 



#### 5.2 Unscheduled Visits

Any visit that occurs between regularly scheduled visits is an Unscheduled Visit. If a subject requires an Unscheduled Visit, he/she must be advised to return to the office wearing the study lenses, if at all possible (unless he/she is experiencing a sign or symptom [as indicated in Section 3.3 Risks and Benefits]). During all unscheduled visits, the Investigator must conduct the following procedures:

- · Assess and record changes in medical condition or concomitant medication
- Assess and record VAs (as applicable)
- Perform biomicroscopy (assessments with or without lenses, as possible)




Status: Effective 

#### · Collect AE and Device Deficiency information

The Investigator may perform additional procedures for proper diagnosis and treatment of the subject. The Investigator must document this information in the subject's case history source documents. If needed, study lenses may be replaced by unmasked site personnel.

If during an Unscheduled Visit the subject is discontinuing the study lenses or discontinuing from the study, the Investigator must conduct Exit procedures according to Table 1-1: Schedule of Study Procedures and Assessments, as possible.

## 5.3 Discontinued Subjects

Discontinued subjects are those who withdraw or are withdrawn from the study after signing the informed consent, including screen failures. Subjects may discontinue from the study at any time for any reason. Subjects may also be discontinued from the study at any time if, in the opinion of the Investigator, their continued participation poses a risk to their health. Discontinued subjects will not be replaced (ie, their subject numbers will not be re-assigned/re-used).

Should a subject exhibit any clinically relevant signs, symptoms, or other clinical observations that possibly could be associated with suspected sensitivity or intolerance to one of the study treatments, the Investigator must document those observations on an AE Form.

Any subject who exits early from the study (excluding screen failures) must undergo all procedures outlined at Visit 4, as applicable.

The Investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, Investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

#### 5.4 Clinical Study Termination

The Study Sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time, for reasonable cause.

If the clinical study is prematurely terminated or suspended by the Study Sponsor:

| Printed By: | Print Date: |
|-------------|-------------|


Status: Effective 

The Study Sponsor must:

- Immediately notify the Investigator(s) and subsequently provide instructions for study termination.
- Inform the Investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension, as applicable.
- The Investigator must:
  - Promptly notify the IRB of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for post-study treatment options as needed.

The Investigator may terminate a site's participation in the study for reasonable cause.

#### 6 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized with counts and percentages from each category. Any deviations to this analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

#### 6.1 Subject Evaluability

The final subject evaluability will be determined prior to breaking the code for masked treatment sequence assignment and locking the database, based on the Deviations and Evaluability Plan.

## 6.2 Analysis Data Sets

#### 6.2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed.


Status: Effective 

## 6.3 Demographic and Baseline Characteristics

Demographic information (age, sex, ethnicity, race) will be summarized on the Safety Analysis Set. Digital fatigue questionnaire collected at Visit 1 will also be summarized on the Safety Analysis Set)

## **6.4 Effectiveness Analyses**

This study defines one primary endpoint, one secondary endpoint

The Safety Analysis Set will serve as the primary set for all effectiveness analyses.

## 6.4.1 Primary Effectiveness

The primary objective of this study is to explore overall vision with BIOFINITY ENERGYS as compared to BIOFINITY lenses after 1 week of wear. The primary endpoint is the subjective rating of overall vision, collected binocularly on a scale of 1 (Poor) to 10 (Excellent).

## 6.4.1.1 Statistical Hypotheses

No inferences are to be made on the primary effectiveness endpoint, therefore no hypotheses are formulated.

## 6.4.1.2 Analysis Methods

Descriptive statistics will be provided.

#### **6.4.2** Secondary Effectiveness

The secondary objective of this study is to evaluate the difference in over-refraction of BIOFINITY ENERGYS as compared to BIOFINITY. The secondary endpoint is the over-refraction, collected in diopters for each eye at Dispense.

#### **6.4.2.1** Statistical Hypotheses

No inferences are to be made on the secondary effectiveness endpoint, therefore no hypotheses are formulated.

## 6.4.2.2 Analysis Methods

Descriptive statistics will be provided.


Status: Effective 



# 6.5 Subgroup Analyses

It is not expected that demographic or baseline characteristics will have an impact on the study results in this study. No subgroup analyses are planned.


Status: Effective 

## 6.6 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for the primary analysis.

## 6.7 Multiplicity

No multiplicity adjustment needs to be considered for the effectiveness endpoints since no formal hypothesis testing will be conducted.

## **6.8** Safety Analysis

The safety endpoints for this study are AEs, biomicroscopy findings, and device deficiencies.

Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation, significant non-serious AEs, and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to study lenses.

Each biomicroscopy parameter will be tabulated by its grade. For each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (Visit 2 or Visit 1, if Visit 2 and Visit 1 occur on the same date) to any subsequent visit will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits for these eyes experiencing the increase.

Two listings (prior to exposure of study lenses and treatment-emergent) of device deficiencies, as recorded on the Device Deficiency Form, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be done for safety analysis.

#### 6.9 Interim Analyses

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.


Status: Effective 

# 6.10 Sample Size Justification

No formal sample size calculation is provided given the pilot and descriptive nature of the study.

## 7 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### **Terms and Definitions**

| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or injury, or |
|---|---|
| | untoward clinical signs (including abnormal laboratory findings) in |
| | subjects, users or other persons, whether or not related to the |
| | investigational medical device (test product). Note: For subjects, |
| | this definition includes events related to the test product, the |
| | control product, or the procedures involved. For users or other |
| | persons, this definition is restricted to events related to the test |
| | product. |
| Adverse Device | AE related to the use of an investigational medical device (test |
| Effect (ADE) | product) or control product. Note: This definition includes AEs |
| | resulting from insufficient or inadequate instructions for use, |
| | deployment, implantation, installation, or operation; any |
| | malfunction; and use error or intentional misuse of the test product |
| | or control product. |
| Anticipated Serious | Serious ADE which by its nature, incidence, severity or outcome |
| Adverse Device | has been identified in the risk management file. |
| Effect (ASADE) | |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, quality, |
| | durability, reliability, safety, or performance. Note: This definition |
| | includes malfunctions, use errors, and inadequate labeling. |
| Malfunction | Failure of a medical device to meet its performance specifications |
| | or otherwise perform as intended. Performance specifications |
| | include all claims made in the labeling of the device. The intended |
| | performance of the device refers to the intended use for which the |
| | device is labeled or marketed. |
| Non-serious Adverse | AE that does not meet the criteria for an SAE. |
| Event | |
| Serious Adverse | AE that led to any of the following: |
| Event (SAE) | Death. |

Effective Date: 01-Mar-2018 Alcon - Business Use Only Protocol - Clinical Effective


Document: TDOC-0054838
Status: Effective 

| A serious deterioration in the health of the subject that either resulted in: a) a life-threatening illness or injury. Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form. b) any potentially sight-threatening event or permanent impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization are diverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non- Serious Adverse Event A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. Unanticipated | | |
|---|---|---|
| a) a life-threatening illness or injury. Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form. b) any potentially sight-threatening event or permanent impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) A significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | A serious deterioration in the health of the subject that either |
| Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form. b) any potentially sight-threatening event or permanent impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | resulted in: |
| immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form. b) any potentially sight-threatening event or permanent impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | a) a life-threatening illness or injury. |
| does not include an event which hypothetically might have caused death had it occurred in a more severe form. b) any potentially sight-threatening event or permanent impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | Note: Life-threatening means that the individual was at |
| caused death had it occurred in a more severe form. b) any potentially sight-threatening event or permanent impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | immediate risk of death from the event as it occurred, ie, it |
| b) any potentially sight-threatening event or permanent impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | does not include an event which hypothetically might have |
| impairment to a body structure or a body function. c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | caused death had it occurred in a more severe form. |
| c) in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | b) any potentially sight-threatening event or permanent |
| Note: Planned hospitalization for a pre-existing condition, without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | impairment to a body structure or a body function. |
| without serious deterioration in health, is not considered an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | <ul> <li>c) in-patient hospitalization or prolonged hospitalization.</li> </ul> |
| an SAE. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | Note: Planned hospitalization for a pre-existing condition, |
| individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non- Serious Adverse Event A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | without serious deterioration in health, is not considered |
| observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | an SAE. In general, hospitalization signifies that the |
| overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | individual remained at the hospital or emergency ward for |
| physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | observation and/or treatment (usually involving an |
| that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | |
| complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | |
| serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | |
| whether "hospitalization" occurred, the event should be considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | complication prolongs hospitalization or fulfills any other |
| considered serious. d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 7.1 for additional SAEs. Serious Adverse Device Effect (SADE) Significant Non- Serious Adverse Possible A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | serious criteria, the event is serious. When in doubt as to |
| d) a medical or surgical intervention to prevent a) or b). e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. **Refer to Section 7.1 for additional SAEs.** Serious Adverse Device Effect (SADE) Significant Non- Serious Adverse Event A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. **Refer to Section 7.1 for additional Significant Non-Serious AEs.** | | whether "hospitalization" occurred, the event should be |
| e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. **Refer to Section 7.1 for additional SAEs.** Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. **Refer to Section 7.1 for additional Significant Non-Serious AEs.** | | |
| test results when used within manufacturer's instructions for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. **Refer to Section 7.1 for additional SAEs.** Serious Adverse Device Effect (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. **Refer to Section 7.1 for additional Significant Non-Serious AEs.** | | d) a medical or surgical intervention to prevent a) or b). |
| for use. • Fetal distress, fetal death, or a congenital abnormality or birth defect. *Refer to Section 7.1 for additional SAEs.* Serious Adverse Device Effect (SADE) Significant Non- Serious Adverse Event A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. *Refer to Section 7.1 for additional Significant Non-Serious AEs.* | | e) any indirect harm as a consequence of incorrect diagnostic |
| Fetal distress, fetal death, or a congenital abnormality or birth defect. *Refer to Section 7.1 for additional SAEs.* Serious Adverse | | test results when used within manufacturer's instructions |
| defect. Refer to Section 7.1 for additional SAEs. Serious Adverse ADE that has resulted in any of the consequences characteristic of an SAE. (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | for use. |
| defect. Refer to Section 7.1 for additional SAEs. Serious Adverse ADE that has resulted in any of the consequences characteristic of an SAE. (SADE) Significant Non-Serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | Fetal distress, fetal death, or a congenital abnormality or birth |
| Serious Adverse Device Effect (SADE) Significant Non- Serious Adverse Event ADE that has resulted in any of the consequences characteristic of an SAE. A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | |
| Device Effect (SADE) Significant Non- Serious Adverse Event A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | | Refer to Section 7.1 for additional SAEs. |
| (SADE) Significant Non- Serious Adverse Event A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | Serious Adverse | |
| Significant Non- Serious Adverse Event A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 7.1 for additional Significant Non-Serious AEs. | Device Effect | an SAE. |
| Serious Adverse non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. *Refer to Section 7.1 for additional Significant Non-Serious AEs.* | (SADE) | |
| Event contact lens wear for greater than or equal to 2 weeks. *Refer to Section 7.1 for additional Significant Non-Serious AEs.* | Significant Non- | A significant non-serious AE is a symptomatic, device-related, |
| Refer to Section 7.1 for additional Significant Non-Serious AEs. | Serious Adverse | non-sight threatening AE that warrants discontinuation of any |
| | Event | contact lens wear for greater than or equal to 2 weeks. |
| Unanticipated Serious adverse device effect which by its nature, incidence, | | Refer to Section 7.1 for additional Significant Non-Serious AEs. |
| | Unanticipated | Serious adverse device effect which by its nature, incidence, |


Status: Effective 

| Serious Adverse | severity or outcome has not been identified in the risk management |
|---|---|
| Device Effect | file. |
| (USADE) | |
| Use Error | Act or omission of an act that results in a different medical device |
| | response than intended by manufacturer or expected by user. |
| | Note: This definition includes slips, lapses, and mistakes. An |
| | unexpected physiological response of the subject does not in itself |
| | constitute a use error. |

## 7.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test *product*).

Figure 7–1 Categorization of All AEs




Status: Effective 

Figure 7-2 Categorization of All Serious Adverse Events



## **Specific Events Relevant to this Protocol**

#### Serious Adverse Events

In addition to reporting all AEs (serious and non-serious) meeting the definitions, the Investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics:
  - o Central or paracentral location
  - o Penetration of Bowman's membrane
  - o Infiltrates > 2 mm diameter
  - o Iritis
  - Increase in intraocular pressure
  - Culture positive for microorganisms
  - o Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon


Status: Effective 

Hyphema

- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting ≥ 50% of corneal surface area

#### Significant Non-Serious Adverse Events

A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. In addition, the Investigator must report any occurrence of the following as a Significant Non-Serious AE:

- Peripheral non-progressive non-infectious ulcers
- All symptomatic corneal infiltrative events
- Corneal staining score greater than or equal to Grade 3 (see CLD523-E001 MOP for grading scales)
- Temporary vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that persists for 2 or more weeks
- Neovascularization score greater than or equal to Grade 2 (see CLD523-E001 MOP for grading scales)

The above events are based upon the categories provided in the ISO 11980 and the US FDA Premarket Notification (510(k)) Guidance Document for Daily Wear Contact Lenses and Contact Lens Care Products.

#### Device Deficiencies

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with patient harm (ie, ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The Investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any patient harm separately. Examples of device deficiencies include the following:

| Printed By: | Print Date: |
|-------------|-------------|


Status: Effective 

 Failure to meet product specifications (eg, incorrect lens power/diameter/base curve/color)

- Lens/solution cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (eg, mislabeled product, tampered seal, leaking bottle/container)
- Suspect product contamination
- · Lack of performance

## 7.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the Investigator should inquire about AEs by asking the standard questions:

- "Have you had any health problems since your last study visit?"
- · "Have there been any changes in the medicines you take since your last study visit?"

Additionally, changes in *any protocol-specific parameters and/or questionnaires* evaluated during the study are to be reviewed by the Investigator. Any untoward (unfavorable and unintended) change in *a protocol-specific parameter or questionnaire response* that is clinically relevant, in the opinion of the Investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

## 7.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any pre-existing medical conditions or signs/symptoms present in a subject prior to the start of the study (ie, before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the Investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.

 ADEs or SAEs are documented on the Serious Adverse Event and Adverse Device Effect eCRF within 24 hours of the Investigator's or site's awareness.


Device deficiencies and decumented on the Device Deficiency of CDF within 24 hours of


 Device deficiencies are documented on the Device Deficiency eCRF within 24 hours of the Investigator's or site's awareness.

- A printed copy of the completed Serious Adverse Event and Adverse Device Effect and/or Device Deficiency eCRF must be included with product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report,
- Certificate of Death, etc, if applicable, in narrative section of the Serious Adverse Event and Adverse Device Effect eCRF.

Note: Should the EDC system become non-operational, the site must complete the appropriate paper Serious Adverse Event and Adverse Device Effect and/or Device Deficiency Form. The completed form is emailed to the Study Sponsor at msus.safety@alcon.com according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.

Study Sponsor representatives may be contacted for any protocol related question.

Further, depending upon the nature of the AE or device deficiency being reported, the Study Sponsor may request copies of applicable portions of the subject's medical records. The Investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.

#### **Intensity and Causality Assessments**

Where appropriate, the Investigator must assess the intensity (severity) of the AE based upon medical judgment with consideration of any subjective symptom(s), as defined below:

#### Intensity (Severity)

Status: Effective

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.


Status: Effective 

Severe An AE is severe if the sign or symptom is incapacitating and results in the subject's inability to work or engage in their usual activities.

For every AE in the study, the Investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by Study Sponsor utilizing the same definitions, as shown below:

#### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (ie, there are other more likely causes for the AE).

The Study Sponsor will assess the AEs and may upgrade the Investigator's assessment of seriousness and/or causality. The Study Sponsor will notify the Investigator of any AEs that are upgraded from non-serious to serious or from unrelated to related.

#### 7.4 Return product analysis

Study lenses associated ONLY with *comfort or vision-related* device deficiencies and/or *comfort or vision related* AEs should be returned and must include a hard copy of the corresponding AE and/or Device Deficiency CRF. These products should be returned to the Sponsor at the end of the study, unless instructed otherwise by the Sponsor.

## 7.5 Follow-Up of Subjects with Adverse Events

The Investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The Investigator should provide the Study Sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of subject exit from study, any additional information received at follow-up should be documented in the eCRFs up to study completion (ie, database lock).


Status: Effective 

Any additional data received up to 1 month after subject discontinuation or exit must be documented and available upon the Study Sponsor's request. All complaints received after this time period will be considered and processed as spontaneous and should be communicated to the medical device's manufacturer as per local requirements.

The Investigator should also report complaints on non-Alcon products directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

## 7.6 Pregnancy in the Clinical Study

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case—by-case basis.

## 8 CONFIDENTIALITY, BIAS, AND MASKING

## 8.1 Subject Confidentiality and Methods Used to Minimize Bias

The Investigator must ensure that the subject's anonymity is maintained throughout the course of the study. In particular, the Investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. At the end of the clinical study, the Sponsor will collect a copy of the enrollment log without any identifying subject information. All documents submitted to the Sponsor will identify the subjects exclusively by number and demographic information. No other personally identifying information should be transmitted to the Sponsor.

This study is double-masked with subjects randomized to use BIOFINITY or BIOFINITY ENERGYS for the duration of the 7 ± 2 day treatment period. The Investigator and Sponsor personnel (other than person responsible for generating the randomization schedule, and unmasked clinical data managers) involved in reporting, obtaining, and/or reviewing the clinical evaluations will be masked to the identity of the contact lens being administered. This level of masking will be maintained throughout the conduct of the study with the exception of the Clinical Project Lead, who may also remain unmasked throughout the study. Unmasking will occur only after all planned study data have been validated, and the database locked. Masked study personnel must avoid seeking information that may compromise masking. Unmasked study personnel must not disseminate information that is potentially unmasking to any masked personnel. The **masked** and **unmasked** site personnel must coordinate all study activities as necessary to protect masking and minimize bias during the trial.


Status: Effective 

## 8.2 Unmasking of the Study Treatment

Masked information on the identity of the assigned medical device should not be disclosed during the study. If the treatment code needs to be broken in the interest of subject safety, the Investigator is encouraged to contact an appropriate Study Sponsor representative prior to unmasking the information if there is sufficient time. Dependent upon the individual circumstances (ie, medical emergency), the code may be broken prior to contact with the Study Sponsor. The Study Sponsor must be informed of all cases in which the code was broken and of the circumstances involved. Additionally, the Study Sponsor may be required to unmask the information in order to fulfill expedited regulatory reporting requirements.

## 9 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

## 9.1 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the eCRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Study monitors are appointed by the Study Sponsor and are independent of study site staff. If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents should include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility
- Date of informed consent
- · Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- · IP accountability records
- Documentation of AEs and other safety parameters (if applicable)
- Records regarding medical histories and the use of concomitant therapies prior to and during the study
- Date of study completion and reason for early discontinuation, if applicable

| Printed By: | Print Date: |
|-------------|-------------|


Status: Effective 

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the eCRF are consistent with the original source data.

Only designated individuals may complete the eCRFs. The eCRFs will be submitted at regular intervals following the clinical study visit schedule. It is expected that all data reported will have corresponding entries in the source documents. The Principal Investigator is responsible for reviewing and certifying that the eCRFs are accurate and complete. The only subject identifiers recorded on the eCRFs will be subject number, and subject demographic information.

#### 9.2 Data Review and Clarifications

Upon completion of the eCRFs, a targeted review of the eCRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. Additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's eCRFs.

## 9.3 Regulatory Documentation and Records Retention

The Investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the Sponsor and the Investigator's files will be reviewed as part of the ongoing study monitoring. Financial disclosure is not subject to regulatory inspection and should be kept separately.

Additionally, the Investigator must keep study records and source documents until the Sponsor provides written approval for their destruction. If the Investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, the Sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations (generally 2 years after discontinuing clinical development or after the last marketing approval).

#### 10 ETHICS AND COMPLIANCE

This trial will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and the referenced directives, regulations, guidelines, and/or standards.


Status: Effective 

## 10.1 Compliance

The Investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The Investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records.

## 10.2 Institutional Review Board (IRB)

This trial requires IRB approval prior to initiation. This protocol, subject informed consent, and subsequent amendments will be reviewed and approved by an IRB.

Before clinical study initiation, this protocol, the ICF (and assent form, if applicable), any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB. The Investigator must provide documentation of the IRB approval to the Study Sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), ICF, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB must be provided with a copy of the Package Insert, any periodic safety updates, and all other information as required by local regulation and/or the IRB. At the end of the study, the Investigator must notify the IRB about the study's completion. The IRB also must be notified if the study is terminated prematurely. Finally, the Investigator must report to the IRB on the progress of the study at intervals stipulated by the IRB.

Voluntary informed consent must be obtained from every subject prior to the initiation of any screening or other study-related procedures. The Investigator must have a defined process for obtaining consent. Specifically, the Investigator, or delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the Investigator, and if required by local regulation, other qualified personnel. The Investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information


Status: Effective 

for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and Sponsor-designated personnel. The Investigator must keep the original, signed copy of the consent and must provide a duplicate copy to each subject according to local regulations. Following this study, the subject will return to their eye care professional for their routine eye care and contact lenses.

## 11 PROTOCOL AMENDMENT HISTORY

| Version | Brief Description and Rationale |
|---|---|
| 1 | Initial Version of this document |
| 2 | Section 1, Page 6 |
| | Exclusion criteria #11 revised: |
| | from |
| | 11. Any use of topical ocular medications and artificial tear or |
| | rewetting drops that would require instillation during contact lens |
| | wear. |
| | to |
| | 11. Any use of topical ocular medications that would require |
| | instillation during contact lens wear. |
| | _ |


Status: Effective 

#### 12 REFERENCES

## 12.1 References applicable for all clinical trials

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- ISO 14155:2011 Clinical investigation of medical devices for human subjects Good clinical practice

## 12.1.1 US references applicable for clinical trials

- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators
- The California Bill of Rights

## 12.2 References for this clinical trial

Not Applicable

Alcon - Business Use Only Protocol - Clinical Effective Document: TDOC-0054838 Version: 2.0; Most-Recent; Effective; CURRENT Status: Effective Effective Date: 01-Mar-2018

| Date/Time<br>(mm/dd/yyyy GMT): | Signed by: | Justification: |
|--------------------------------|------------|----------------|
| 02/28/2018 12:20:36 | | |
| 02/28/2018 20:03:36 | | |
| 03/01/2018 00:28:55 | | |